CLINICAL TRIAL: NCT07322367
Title: A Pragmatic Randomized-Controlled Learning Health System Trial
Brief Title: A Mobile Patient Health Technology Intervention for Improving Lung Cancer Screening Rates in Eligible High Risk Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IRB00139213; P30CA012197 (NIH)
Record Dates: First submitted 2026-01-05; First posted 2026-01-07 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A (Experimental): Patient portal message first followed by up to 3 reminder text messages.
  Interventions: Other: Portal Message with Reminder Text Messages
- Arm B (Experimental): Text message only with up to 3 reminder text messages.
  Interventions: Other: Text Message with Reminder Text Messages
- Arm C (Experimental): Portal message only with no reminder messages.
  Interventions: Other: Portal message only
- Usual Care Arm (Active Comparator): Patients receive usual care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Portal Message with Reminder Text Messages — If the participant has an upcoming scheduled appointment, they will receive a reminder text message 5 days after initial portal message, a final reminder text message a day before their scheduled appointment, and potentially an 'in progress' text message reminder if they start the mPATH-Lung program but do not complete it.
  If the participant does not have an upcoming scheduled appointment, they will receive a reminder text message 5 days after initial portal message, the final reminder message 8 days after the initial message, and potentially an 'in progress' text message reminder.
  Arms: Arm A
Other: Text Message with Reminder Text Messages — If the participant has an upcoming scheduled appointment, they will receive a reminder text message 5 days after initial message, a final reminder text message a day before their scheduled appointment, and potentially an 'in progress' text message reminder.
  If the participant does not have an upcoming scheduled appointment, they will receive a reminder text message 5 days after initial message, the final reminder message 8 days after the initial message, and potentially an 'in progress' text message reminder.
  Arms: Arm B
Other: Portal message only — Participant will only receive portal message with no reminder text messages.
  Arms: Arm C
Other: Usual Care — Standard of care
  Arms: Usual Care Arm

SUMMARY:
To evaluate the real-world effectiveness and implementation strategies for mPATH-Lung, investigators propose a pragmatic, randomized controlled trial across an academic Learning Health System. The trial will contrast several approaches to participant outreach and will specifically target engaging fully powered cohorts of racial/ethnic minorities and rural residents.

DETAILED DESCRIPTION:
Primary Objective: Evaluate the real-world effectiveness of mPATH-Lung in increasing lung cancer screening rates across diverse populations.

Secondary Objectives

* Compare the differential effectiveness of three outreach strategies for engaging participants with mPATH-Lung across vulnerable rural or ethnic/racial minority population subgroups.
* Estimate the additional revenue generated by mPATH-Lung through increased screening and downstream care.
* Evaluate the potential for over-screening and the impact of applying HEDIS-based exclusion criteria

ELIGIBILITY:
Inclusion Criteria:

Eligible patients will:

* Meet the Medicare criteria for lung cancer screening, as updated in February 2022:
* Age 50 - 77 years
* Smoked at least 20 pack years
* Current smoker or quit smoking within the past 15 years
* Be established with a primary care provider within the Atrium Health Wake Forest Baptist health network (defined as having completed at least 1 primary care appointment in the past 6 months or have completed at least 2 primary care appointments within the past 18 months or being scheduled to see a health network primary care provider within the next 30 days).
* Have a patient portal account or cellphone number listed in the electronic health record
* Have a North Carolina address listed in the electronic health record

Exclusion Criteria:

The following patients will be excluded:

* Patients flagged as needing a language interpreter in the electronic health record for any language other than Spanish (electronic messages and intervention are deliverable in English or Spanish only)
* Those for whom lung cancer screening would be or may be inappropriate:

electronic health record Prior history of lung cancer electronic health record Chest CT within the last 12 months electronic health record Those meeting the HEDIS COL-E measure exclusion criteria based on significant comorbidities and/or frailty.

Ages: 50 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27000 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants to Complete Lung Screening CT - Primary Effectiveness | 90 days
  Completion of the lung screening CT by participants.

SECONDARY OUTCOMES:
Number of Participants with Eligibility for Lung Screening | 90 days
  Reach of the mPATH-Lung platform, defined as the participants who determine their eligibility for lung screening within the mPATH-Lung program within 90 days of the first invitation. Investigators will determine reach overall, within subgroups, and within study arms.
Number of Requests for Lung Screening | 90 days
  Requests for lung screening within the mPATH-Lung program
Number of Orders for Lung Screening CT Scans | Within 90 days of randomization
  Orders for lung screening CT scans for participants in study arms
Amount of Revenue Generated | 12 months following completion of screenings
  Revenue (costs) generated from lung cancer screening and follow-up care.
Number of Participants that Represent Over-screening | 90 days
  Among patients with newly diagnosed lung cancer by lung screening, the participants that represent over-screening, defined as a patient being deemed too ill for potentially curative surgery on blinded chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Brent Heideman, Jr., MD, Principal Investigator — Wake Forest Baptist Comprehensive Cancer Center
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No